CLINICAL TRIAL: NCT06860802
Title: Aim 3 - Precision Coordination of Therapeutic and Prophylactic Antibiotics to Reduce Infection, Toxicity, and Emergence of Resistance Following Acute Abdominal Surgery
Brief Title: Precision Antibiotic Dosing for Appendectomy
Acronym: PANDA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manjunath Prakash Pai, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00263447; R01HS027788 (AHRQ)
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Appendicitis (Diagnosis)
Keywords: Cefoxitin; Appendectomy; Surgical Site Infections
MeSH Terms: conditions — Appendicitis; Disease; Surgical Wound Infection | interventions — Cefoxitin

STUDY DESIGN:
Intervention Model Description: This is an interventional phase 1 study design that includes human adult participants undergoing an appendectomy. The study entails collection and analysis of three blood (plasma) samples, two subcutaneous fat samples, and appendix tissue samples from resected surgical specimens. The intervention is to receive the standard of care surgical prophylaxis or the standard of care surgical prophylaxis plus the addition of cefoxitin 2000 mg within 30 minutes of incision
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): The current standard of care surgical prophylaxis regimen
- Cefoxitin (Experimental): Administration of Cefoxitin 2000 mg within 30 minutes of incision to the existing standard of care intervention
  Interventions: Drug: Cefoxitin

INTERVENTIONS:
Drug: Cefoxitin — Cefoxitin 2000 mg Bolus Injection
  Arms: Cefoxitin

SUMMARY:
This research is studying a drug called cefoxitin already approved by the Food and Drug Administration (FDA) to reduce the risk of infection after surgery to remove an appendix. Researchers are studying a large group of people to continue to learn how best to dose antibiotics. This research will compare the current standard treatment which is a single dose prior to surgery to a new method that includes adding another dose of cefoxitin within 30 minutes of starting the surgery. This study will measure cefoxitin concentrations in blood, fat, and appendix tissue samples to compare the standard dosing method to our new method. This information will help us figure out the right dose of this drug to prevent infection after surgery to remove an appendix.

DETAILED DESCRIPTION:
This interventional, phase 1 study aims to improve surgical site infection (SSI) prevention in patients undergoing appendectomy for uncomplicated appendicitis. Despite standard antibiotic prophylaxis, SSI rates remain high, with a pelvic abscess risk of 9.4%. Current prophylactic antibiotic regimens may not achieve optimal tissue concentrations, especially in fat and appendix tissue.

This study will evaluate the probability of target attainment (PTA) of cefoxitin, cefuroxime, and metronidazole in plasma, subcutaneous fat, and appendix tissue. A cohort of 46 adult patients will be randomized to receive standard-of-care antibiotics with or without an additional cefoxitin dose. Antibiotic concentrations will be measured in collected blood, fat, and appendix samples.

The study's primary objective is to determine whether a supplemental cefoxitin dose improves PTA compared to standard prophylaxis. Population pharmacokinetic modeling will validate the intervention's effectiveness in optimizing antibiotic exposure and reducing SSI risk. The results may inform future precision antibiotic dosing strategies for appendectomy and other acute care surgeries.

Primary Outcome Measure:

Probability of achieving 50% time above 8 mcg/mL (cefuroxime or cefoxitin) in appendix tissue between intervention and standard care groups.

Study Design:

Randomized, interventional, phase 1 study Enrollment: 46 participants Inclusion: Adults (>18 years) undergoing appendectomy for acute appendicitis Exclusion: Pregnant individuals, prisoners, patients with perforation or abscess This study seeks to improve perioperative antibiotic management, reducing SSI rates while minimizing unnecessary antibiotic exposure and resistance development.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute appendicitis and plan to undergo appendectomy at the University of Michigan

Exclusion Criteria:

* Prisoners
* Patients that are pregnant
* Patients with perforation or abscess on CT Scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Probability of Achieving Optimal Antibiotic Concentration in Appendix Tissue | 4 hours
  The probability of achieving 50% time above 8 mcg/mL (cefuroxime or cefoxitin) in appendix tissue in the intervention compared to the non-intervention (standard of care) arm.

CONTACTS AND LOCATIONS:
Overall Officials: Manjunath Pai, PharmD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT06860802/ICF_000.pdf